CLINICAL TRIAL: NCT01749150
Title: STUDY TO EVALUATE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND ANTIVIRAL ACTIVITY OF RITONAVIR-BOOSTED DANOPREVIR IN COMBINATION WITH PEGINTERFERON ALFA-2A PLUS RIBAVIRIN IN TREATMENT-NAÏVE PATIENTS OF ASIAN ORIGIN WHO HAVE CHRONIC HEPATITIS C GENOTYPE 1 WITH OR WITHOUT COMPENSATED CIRRHOSIS
Brief Title: A Study of Ritonavir-Boosted Danoprevir in Combination With Pegasys (Peginterferon Alfa-2a) and Copegus (Ribavirin) in Patients of Asian Origin With Chronic Hepatitis C Genotype 1 With or Without Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YV28218
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — danoprevir; Ritonavir; peginterferon alfa-2a; Ribavirin

ARMS (2):
- with cirrhosis (Experimental)
  Interventions: Drug: danoprevir + ritonavir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]
- without cirrhosis (Experimental)
  Interventions: Drug: danoprevir + ritonavir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]

INTERVENTIONS:
Drug: danoprevir + ritonavir — 125 mg danoprevir + 100 mg ritonvir fixed-dose combination tablet, orally b.i.d., 12 weeks
  Arms: without cirrhosis
Drug: danoprevir + ritonavir — 125 mg danoprevir + 100 mg ritonvir fixed-dose combination tablet, orally b.i.d., 24 weeks
  Arms: with cirrhosis
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc weekly, 12 weeks
  Arms: without cirrhosis
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc weekly, 24 weeks
  Arms: with cirrhosis
Drug: ribavirin [Copegus] — 1000-1200 mg orally daily in divided doses, 12 weeks
  Arms: without cirrhosis
Drug: ribavirin [Copegus] — 1000-1200 mg orally daily in divided doses, 24 weeks
  Arms: with cirrhosis

SUMMARY:
This Phase II, open-label, parallel-arm study will evaluate the safety, tolerability, pharmacokinetics and antiviral activity of ritonavir-boosted danoprevir in combination with Pegasys (peginterferon alfa-2a) and Copegus (ribavirin) in treatment-naïve patients of Asian origin with chronic hepatitis C genotype 1. Patients will receive danoprevir 125 mg plus ritonavir 100 mg as fixed dose tablet orally twice daily in combination with weekly Pegasys 180 mcg subcutaneously and Copegus 1000-1200 mg orally daily in divided doses. Treatment duration is 12 weeks in patients without cirrhosis and 24 weeks in patients with compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of East Asian or Southeast Asian origin, >/= 18 years of age
* Presence of chronic genotype 1 hepatitis C infection
* Treatment-naïve

Exclusion Criteria:

* History or presence of decompensated liver disease
* Presence or history of non-hepatitis C chronic liver disease
* Positive for hepatitis B or HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 1.5 years
Pharmacokinetics: Area under the concentration-time curve (AUC) for danoprevir/ritonavir | up to 14 days
Antiviral activity: Change in HCV RNA levels, measured using Roche COBAS TaqMan HCV Test v2.0 for High Pure System | from baseline to Week 36/48
Antiviral activity: Proportion of patients with unquantifiable/undetectable HCV RNA during the study | approximately 1.5 years

SECONDARY OUTCOMES:
Incidence of viral resistance to danoprevir | approximately 1.5 years
Rapid virological response (RVR): Proportion of patients with undetectable HCV RNA at Week 4 | approximately 1.5 years
Complete early virological response (cEVR): Proportion of patients with undetectable HCV RNA at Week 12 | approximately 1.5 years
Sustained virological response 12 weeks after end of treatment (SVR-12), defined as unquantifiable HCV RNA 8-20 weeks after the last day of study drug administration | approximately 1.5 years
Sustained virological response 24 weeks after end of treatment (SVR-24), defined as unquantifiable HCV RNA > 20 weeks after the last day of study drug administration | approximately 1.5 years
SVR measured as HCV RNA log10 IU/mL change from baseline to Week 12 | approximately 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- South Korea (2):
  - Busan
  - Seoul
- Taiwan (6):
  - Chiayi County
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
  - Yunlin County
- Thailand (2):
  - Bangkok
  - Chiang Mai